CLINICAL TRIAL: NCT00659048
Title: Investigation of Potential Additive Inhibitory Effects on HPA-Axis of Ciclesonide Nasal Spray When Administered Concomitantly With Orally Inhaled Beclomethasone Dipropionate (HFA-BDP) in Patients (18-60 Years) With Perennial Allergic Rhinitis (PAR)
Brief Title: Investigation of Potential Additive Inhibitory Effects on HPA-Axis of Ciclesonide Nasal Spray When Administered Concomitantly With Orally Inhaled Beclomethasone Dipropionate (HFA-BDP) in Patients With Perennial Allergic Rhinitis (PAR) (BY9010/M1-408)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-408
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial Allergic Rhinitis; Ciclesonide; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Ciclesonide 200µg
  Interventions: Drug: Ciclesonide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — Ciclesonide 200µg versus Placebo
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The primary objective of this study is to demonstrate that there are no clinically relevant additive inhibitory effects on the HPA-axis when ciclesonide nasal spray is concomitantly administered with orally inhaled HFA-BDP. The secondary objectives are to evaluate safety and tolerability of the combined dosing regimen of orally inhaled HFA-BDP and ciclesonide nasal spray.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 - 60 years of age.
2. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial.
3. A history of PAR for a minimum of one year immediately preceding the Screening Visit.
4. A demonstrated sensitivity to at least one allergen known to induce PAR through a standard prick or intradermal test. A positive test is defined as a wheal diameter at least 3 mm larger than the control wheal for the prick test, and 7 mm or greater than the control for the intradermal test. Documentation of a positive result within 12 months prior to the Screening Visit is acceptable.
5. Females of child-bearing potential are currently taking and will continue to use a medically reliable method of contraception for the entire study duration (e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection). Women of childbearing potential, or less than 1 year postmenopausal, will require a negative plasma pregnancy test at the Screening Visit as well as at last on-treatment visit.
6. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and compliance with all study requirements (visits, record keeping, etc).
7. Normal body weight as evidenced by a Body Mass Index (BMI) between ³ 18 and 31 kg/m², and a body weight > 45 kg.

Exclusion Criteria:

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the study period.
2. History or physical findings of nasal pathology, including nasal polyps (within the last 60 days) or other clinically significant respiratory tract malformations, recent nasal biopsy (within the last 60 days), nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days).
3. Participation in any investigational drug trial within the 30 days preceding the Screening Visit (S0).
4. A known hypersensitivity to any corticosteroid or any of the excipients in the formulations.
5. History or current evidence of clinically relevant allergies or idiosyncrasy to drugs or food.
6. History of alcohol or drug abuse within the preceding two years.
7. History of a positive test for HIV, hepatitis B or hepatitis C.
8. Use of any prohibited concomitant medications within the prescribed (per protocol) withdrawal periods prior to the Screening Visit (S0) and during entire study duration.
9. Previous participation in an intranasal ciclesonide study.
10. Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit (S0).
11. Exposure to corticosteroids for any indication, chronic or intermittent (e.g.: asthma, contact dermatitis), during the past 2 months, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
12. Use of topical corticosteroids in concentrations in excess of the equivalent of 1% hydrocortisone for dermatological conditions during the past 1 month, or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study.
13. Clinically relevant abnormalities in clinical chemical, hematological or any other laboratory variables.
14. Chronic or clinically relevant acute infections.
15. Vegetarian diet or other unusual dietary habits that would preclude the subject's acceptance of standardized meals.
16. Blood donation within the last 30 days before start of the study.
17. Patients that do not have regular sleep patterns (e.g. working at night and sleeping during the daylight hours).
18. Active asthma requiring treatment with inhaled or systemic corticosteroids; intermittent use of beta agonists is acceptable.
19. History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, the common cold, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit (S0), or development of a respiratory infection during the Run-in Period.
20. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (S0). Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit (S0) AND is expected to continue throughout the trial.
21. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit (S0) AND use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
22. Failure to adequately understand and comply with the HFA-BDP instructions or failure to properly administer study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2004-12; Primary Completion 2005-04 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
24 h plasma cortisol profiles and urinary cortisol | 53 days

SECONDARY OUTCOMES:
24-hour urinary cortisol will be monitored at the following times | 53 days
Adverse events | 53 days
vital signs | 53 days

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana/Nycomed, San Antonio, Texas, United States

REFERENCES:
- See also: BY9010-M1-408-RDS-2005-12-05.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4536&filename=BY9010-M1-408-RDS-2005-12-05.pdf